CLINICAL TRIAL: NCT00103116
Title: Autologous Dendritic Cell Vaccines in Non-small Cell Lung Cancer (NSCLC)
Brief Title: Vaccine Therapy in Treating Patients With Stage I, Stage II, or Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edward Hirschowitz (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Edward Hirschowitz, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000410830; R21CA091624 (NIH); UKMC-IRB-0391-F2R (Other: IRB); UKMC-CTRF-G-01-009 (Other Grant/Funding Number: Cancer Treatment Research Foundation)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous dendritic cell cancer vaccine (Experimental): Open label nonrandomized
  Interventions: Biological: autologous dendritic cell cancer vaccine

INTERVENTIONS:
Biological: autologous dendritic cell cancer vaccine — Dendritic cells made from white blood cells obtained through out-patient leukapheresis procedure.
  Vaccine given by injection under the skin in the front, upper thigh. Two vaccine injections total, given one month a part.
  Other Names: DC vaccine; autologous DC vaccine

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells and allogeneic tumor cells may make the body build an effective immune response to kill tumor cells.

PURPOSE: This phase II trial is studying how well vaccine therapy works in treating patients with stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the immunologic effects of adjuvant vaccine therapy comprising autologous dendritic cells loaded with allogeneic non-small cell lung cancer (NSCLC) cells in patients with unresectable stage IIIA or IIIB, or resected stage I-IIIB NSCLC.
* Determine the potential clinical efficacy of this vaccine in these patients.

OUTLINE: This is an open-label study. Patients are stratified according to type of prior primary therapy (surgical vs nonsurgical).

Patients undergo leukapheresis over 3-4 hours to harvest mononuclear cells for the production of dendritic cells (DC). DC are then pulsed with allogeneic non-small cell lung cancer cells to produce an autologous dendritic cell vaccine. Patients receive vaccine intradermally once a month for 2 months in the absence of disease recurrence or unacceptable toxicity.

Patients are followed monthly for 4 months, every 6 months for 2 years, and then periodically thereafter.

PROJECTED ACCRUAL: A total of 60 patients (30 per stratum) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC)

  * Meets 1 of the following stage criteria:

    * Completely resected stage I-IIIB disease

      * Underwent surgical resection > 4 weeks but ≤ 4 years ago
    * Unresectable stage IIIA or IIIB disease AND previously treated with definitive radiotherapy or chemotherapy > 6 weeks ago
  * Bronchoalveolar carcinomas allowed
* Clinically stable disease by chest x-ray or CT scan within the past 6 weeks

  * No progressive disease
* No malignant pleural or pericardial effusions

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ 9.0 g/dL

Hepatic

* Bilirubin ≤ 2.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* No known history of infectious hepatitis

Renal

* Creatinine ≤ 3 mg/dL
* Ionized calcium ≥ 0.9 mmol/L (may be replaced)

Cardiovascular

* No known New York Heart Association class III-IV congestive heart failure
* No hemodynamically significant valvular heart disease
* No myocardial infarction within the past 6 months
* No active angina pectoris
* No uncontrolled ventricular arrhythmia
* No stroke within the past year
* No known cerebrovascular disease
* No other significant cardiac disease by echocardiogram, stress test, or risk assessment by cardiologist (for patients suspected of cardiac disease by history or physical exam)

Immunologic

* No known HIV positivity
* No other immunosuppressive disorders, including chronic disorders

Other

* Not pregnant
* Negative pregnancy test
* Potassium ≥ 3.0 mEq/L (may be replaced)
* Able to tolerate modest blood volume and electrolyte shifts during leukapheresis
* No other malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior biologic therapy allowed
* Other concurrent biologic therapy allowed

Chemotherapy

* See Disease Characteristics
* No concurrent chemotherapy

Endocrine therapy

* No concurrent steroids during and for 16 weeks after study treatment

Radiotherapy

* See Disease Characteristics
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* Prior neoadjuvant or adjuvant therapy for surgically resected patients allowed
* No concurrent shorter courses of immunosuppressive medications during and for 16 weeks after study treatment
* No concurrent chronic immunosuppressive medications
* Concurrent cyclooxygenase-2 inhibitors allowed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Hirschowitz, MD, Study Chair — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky, United States

REFERENCES:
- [Result] Hirschowitz EA, Foody T, Hidalgo GE, Yannelli JR. Immunization of NSCLC patients with antigen-pulsed immature autologous dendritic cells. Lung Cancer. 2007 Sep;57(3):365-72. doi: 10.1016/j.lungcan.2007.04.002. Epub 2007 May 16. PMID 17509725
- [Result] Hirschowitz EA, Foody T, Kryscio R, Dickson L, Sturgill J, Yannelli J. Autologous dendritic cell vaccines for non-small-cell lung cancer. J Clin Oncol. 2004 Jul 15;22(14):2808-15. doi: 10.1200/JCO.2004.01.074. PMID 15254048
- [Result] Hirschowitz EA, Yannelli JR. Immunotherapy for lung cancer. Proc Am Thorac Soc. 2009 Apr 15;6(2):224-32. doi: 10.1513/pats.200806-048LC. PMID 19349492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-randomized open label; stage I-IIIB NSCLC. Closed to accrual in 2006 when defined phase I immunological endpoints were reached.
Pre-assignment Details: None excluded; all completed.
Groups:
- Vaccine: therapeutic autologous dendritic cells : Dendritic cells made from white blood cells obtained through out-patient leukapheresis procedure. Vaccine given by injection under the skin in the front, upper thigh. Two vaccine injections total, given one month a part.
Period: Overall Study
Arm/Group | Vaccine
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 31
  Israel | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Showing Immunologic Response to Vaccine Within Six Months of Immunization
Description: Antigen specific reaction is measured serially in blood of each participant prior to and through six months post-vaccine. Increase in levels of specific T cell activity from pre vaccine to post vaccine serve as primary measures of an individual's response to vaccine. The number (relative percent) of participants achieving immunologic response to vaccine within 6 month of immunization was the dominant metric of vaccine activity within the study population.
Time Frame: six months post vaccine
Measure: Number; unit: participants with immunological response
Arm/Group | Vaccine
Number analyzed (Participants) | 32
participants with immunological response | 22

2. Secondary Outcome: Number of Participants Alive Five Years Post Vaccine
Description: Documentation of radiographic surveillance for recurrence or progression for 5 years post-vaccine
Time Frame: five years post vaccine
Measure: Number; unit: participants
Arm/Group | Vaccine
Number analyzed (Participants) | 32
participants | 20

ADVERSE EVENTS:
Time Frame: five years
Arm/Group | Vaccine
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 16/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=32)
injection site reaction (General disorders) | 16 (16) — Self limited injection site reaction was observed in half the study participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No